CLINICAL TRIAL: NCT03731728
Title: The Effectiveness of Group CBT and Exercise in Management of Depression: A Three Arm Randomized Controlled Pilot Trial
Brief Title: Group CBT and Exercise in Management of Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00080975
Record Dates: First submitted 2018-10-21; First posted 2018-11-06 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the database which contains the randomization code. In addition, study participants will self-complete all outcome assessments on a tablet with the assessor only guiding the process. Moreover, these assessors will not be involved in data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group CBT plus TAU (Experimental): Participants enrolled in the "group CBT plus TAU" arm of the study will receive a 2-hour session of group CBT every week for 14 weeks in addition to being wait-listed to receive treatment as usual.
  Interventions: Behavioral: Group CBT
- Group Exercise plus TAU (Experimental): Participants enrolled in the "group exercise plus TAU" arm of the study will receive 50 minutes of scheduled and facilitated exercises three times a week for 14 weeks in addition to being wait-listed to receive treatment as usual.
  Interventions: Behavioral: Group exercise
- Wait-listing for TAU (No Intervention): Participants enrolled in the wait-listing for "treatment as usual" or TAU arm of the study will be wait-listed to receive individual therapy or counselling from an Addiction and Mental Health therapist as per current standard protocol for managing patients with MDD at Addiction and Mental Health Clinics of Edmonton Zone.

INTERVENTIONS:
Behavioral: Group CBT — All therapists will use a manualized Cognitive-Behavior Therapy (CBT) protocol with the same handouts and schedule developed based on the book "Mind Over Mood". Group CBT will be provided to a group of maximum 10 participants. Each session will be 2 hours long and will be provided by certified therapists with special training to deliver group CBT. The structure of the session will be agenda setting, check-in, review of homework, new concepts/skills, homework assignment, and feedback.
  Arms: Group CBT plus TAU
Behavioral: Group exercise — Participants enrolled in the group exercise plus TAU arm of the study will be wait-listed for TAU and will receive 50 minutes of scheduled and facilitated exercises three times a week for 14 weeks.
  Arms: Group Exercise plus TAU

SUMMARY:
INTRODUCTION: There is strong evidence indicating the effectiveness of Cognitive-Behavior Therapy (CBT) in the management of Major Depressive Disorder (MDD) and some clinical trials indicating physical exercise (PE) as an effective treatment for the disorder. However, few studies have evaluated the effect of group CBT or PE compared to wait-listing to receive treatment as usual (TAU) in the management of MDD. This study will evaluate and compare the effectiveness of: 1) group CBT plus wait-listing for TAU; versus 2) group PE plus wait-listing for TAU; versus 3) only wait-listing for TAU in management of MDD. The investigators hypothesize that participants with MDD assigned to the group CBT or PE (plus wait-listed for TAU) arms of the study will achieve superior outcomes compared to participants only wait-listed for TAU.

METHODS AND ANALYSIS: This is a prospective rater-blinded randomized controlled trial assessing the benefits for participants with MDD. 120 patients with MDD referred to Addiction and Mental Health (AMH) clinics in Edmonton Zone who are informed about the study and consent to participate will be randomly assigned to one of the 3 arms of the study: 1) 40 participants wait-listed for TAU will receive weekly sessions of group CBT for 14 weeks; 2) 40 participants wait-listed for TAU will receive PE 3 times a week for 14 weeks; and 3) 40 participants will only be wait-listed for TAU. Participants will be assessed at enrollment, 3 and 6 months post enrolment, mid-treatment, and at treatment completion . Their assessments will cover primary outcomes including functional variables (relationships, well-being, physical activity) and symptom variables (changes in depressive symptoms scores). Secondary client outcomes will be service variables (e.g. patient compliance, retention in treatment, patient satisfaction). In addition, participants in the intervention groups will be evaluated weekly with one functional measure. The data will be analyzed using repeated measures and effect size analyses, and correlational analyses will be completed between measures at each time point.

ETHICS AND DISSEMINATION: The study will be conducted in accordance with the Declaration of Helsinki (Hong Kong Amendment) and Good Clinical Practice (Canadian Guidelines). Written informed consent will be obtained from each subject. The study has received ethical clearance from Health Ethics Research Board of the University of Alberta (Ref. # Pro 00080975) and operational approval from the provincial health authority (AHS # 43638). The results will be disseminated at several levels, including patients, practitioners, academics/researchers, and healthcare organizations.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE: Depression with a global prevalence of over 4% is a major public health problem and is the single largest contributor to non-fatal health loss. There is a need to identify interventions that are relatively cost-efficient, scalable, and can be offered to many people. Treatment for depressive disorders typically includes anti-depressant medication and/or counselling and psychotherapy.

Exercise as a form of treatment for depressive disorders, especially of mild-to-moderate severity, has evidence of benefit. In fact, the magnitude of the effect of exercise as a treatment for depression is reported to be comparable to conventional treatment. An umbrella review of systematic reviews and meta-analyses of the use of exercise to treat depressive symptoms in older adults, for example, concluded that exercise is safe and efficacious in reducing depressive symptoms in older people and it should be considered as a core intervention in the multidisciplinary treatment of depression in this age group. A meta-analysis adjusting for publication bias, concluded that "exercise has a large and significant antidepressant effect in people with depression". The mechanisms by which exercise decreases depressive symptoms may include biological mechanisms, such as anti-inflammatory effects or increasing neurotransmitter levels implicated in depression. Other mechanisms may include increasing self-efficacy or enhancing social interaction.

Despite this strong evidence base, few studies have incorporated multiple treatment conditions in a randomized controlled trial design, and few studies appear to have assessed the effect of group CBT. In addition, few studies could be found that compared group CBT, group exercise, and wait-listing for treatment as usual conditions. This is important in further delineating the effective components of treatment for mild to moderate depression, and results have implications for service delivery and clinical recommendations in the treatment of depression within healthcare organizations in Alberta and beyond. Specifically, patients with MDD referred to Addiction and Mental Health (AMH) Clinics in Edmonton Zone may wait for weeks before receiving individual treatment. Thus, if found to be effective, group treatment conditions examined in this study may serve as an expedient treatment avenue to decrease wait-list times for patients with MDD.

AIM AND OBJECTIVES: The aim of the project is to conduct a three-arm randomized controlled pilot trial to evaluate the feasibility and initial efficacy of group CBT or group exercise on depression symptom scores and quality of life measures in patients with MDD. The client outcomes will be organized according to: functional variables (relationships, well-being, physical activity), symptom variables (change in depressive symptoms scores), and service variables (e.g. patient compliance and retention in treatment and patient satisfaction).

Given the aim, the objectives of the project are to compare mean changes in functioning, clinical symptoms, and service satisfaction variables from enrolment baseline to 12 weeks post enrolment for: 1) participants receiving group CBT plus wait-listed to receive TAU; 2) participants receiving scheduled exercise plus wait-listed to receive TAU; and 3) those only wait-listed to receive TAU. Another objective of the study is to compare mean changes in functioning, clinical symptoms, and service satisfaction variables from treatment baseline to 7 and 14 weeks post-treatment commencement for: 1) participants receiving group CBT plus wait-listed to receive TAU and 2) participants receiving scheduled exercise plus wait-listed to receive TAU.

HYPOTHESIS: The investigators hypothesize that participants enrolled in the group CBT or group exercise treatments while wait-listed to receive TAU will achieve statistically superior outcomes at 12 weeks post enrollment compared to participants only wait-listed to receive TAU on each outcome measure used. We expect that participants enrolled in group CBT plus TAU will have comparable outcomes to those enrolled in the group exercise plus TAU arm of the study at 7and 14 weeks post treatment commencement.

MATERIALS AND METHODS: This study will be a longitudinal, prospective, parallel design, three-arm, rater-blinded randomized clinical trial with a recruitment period of six months and an observation period of 14 weeks for each participant.

The research will be carried out in a municipal recreational centre as well as AMH clinics in Edmonton, a large, socio-demographically diverse city in Western Canada. Potential participants will be recruited from the AMH Intake Clinic in Edmonton. Patients with depression at intake assessment who are presumed to meet the inclusion criteria of the study will be invited to enroll in this study.

To confirm the diagnosis of MDD using the DSM 5 criteria, potential participants will be sent to the Mood and Anxiety clinic or Urgent Clinics in Edmonton where they will be assessed by one of a group of psychiatrists or psychiatry residents who are independent from the study team. The psychiatrist or resident may or may not initiate, continue or adjust pharmacotherapy. The diagnosis will be communicated to the study coordinator and clinic nurse. The participants with MDD will be informed of their eligibility to participate in the study and will be considered for randomization after providing informed consent whereas patients with other diagnoses will be informed of their exclusion from the study and will be directed to receive an appropriate treatment for their condition.

After diagnostic confirmation by a psychiatrist, a research assistant who is trained in study procedures will provide the potential participants with an information leaflet about the study and answer any related questions they may have. All potential participants who agree to take part in the study will provide written informed consent prior the completion of baseline assessment measures and randomization.

At baseline, demographic and contact information will be collected. The participants' name and contact information will also be collected but only used for future communication or for arrangement of treatment, assessment and follow-up sessions.

Participant's Medical Record will also be reviewed at two points, at the time of enrollment in the study and 6 months after enrollment, to gather information about the participant's use of health services in the past 6 months to compare service utilization among the groups and determine if participation in the intervention group impacts the use of other health services in the short term. This same data can also be used for any economic analyses (i.e., cost-effectiveness) that will be conducted.

All the data will be stored for a minimum of 7 years prior to destruction as per the research ethics board requirements, and research ethics board requirements pertaining to collection and storage of information will be followed.

SAMPLE SIZE: As this is a pilot study, the research will utilize data that can be elicited from participants who can be enrolled within existing operational resources and time frames. The study will therefore be limited to a sample size of 120, with about 40 patients recruited into each arm of the study.

RANDOMIZATION AND BLINDING: Randomization will be enacted via randomly generated codes. Each study participant will receive a randomization code. Because it will not be possible for participants to be blinded, treatment allocation will be made explicit to them as soon as randomization is concluded. Outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the database that contains the randomization code. In addition, study participants will self-complete all outcome assessments with the assessor facilitating procedural aspects if needed. Moreover, these assessors will not be involved in data analysis. After data collection is complete all data will undergo a blind review for the purposes of finalizing the planned analysis.

FOLLOW UP ASSESSMENT: 12 and 24 weeks after baseline assessments, a blinded researcher will contact study participants in all three arms of the study and assist them in the completion of a range of assessment tools related to the outcome measures. The number of treatment sessions (group CBT, group exercise or individual therapy) participants have received at each time point would be recorded for participants in all treatment arms. In addition, participants in the group CBT and exercise arms of the study would complete assessments tools weekly during the sessions and also at mid-treatment (7 weeks after starting treatment) and at the end of the treatment (14 weeks after the treatment commencement). These self-rated assessments would be coordinated by the group facilitators.

STATISTICAL METHODS: The primary goal of the statistical analysis will be to produce summary descriptive statistics for the longitudinal data, which will provide estimates for future sample size calculations and enable calculation of effect size. For the three arm trial, we will compare mean change scores for primary and secondary outcome measures from enrollment baseline to 12 weeks and 24 weeks post-enrollment into the study, whilst for the two arm trial, we will compare mean changes scores for primary and secondary outcome measures from treatment baseline to 7 and 14 weeks post-enrollment into treatment in addition to comparing trends in weekly change scores on the CORE-10 OM between the two intervention groups. The data will be analyzed using repeated measures and effect size analyses, and correlational analyses will be completed between measures at each time point. The results of this study will guide the design for a future, more highly powered, study.

PATIENT AND PUBLIC INVOLVEMENT: The study was designed and finalized based on feedback from patient representatives. This randomized trial also offers patients the opportunity to provide feedback via the patient satisfaction survey.

ETHICS AND DISSEMINATION: The study will be conducted in accordance with the Declaration of Helsinki (Hong Kong Amendment) and Good Clinical Practice (Canadian Guidelines). Written informed consent will be obtained from each participant. The study has received ethical clearance from Health Ethics Research Board of the University of Alberta (Ref. # Pro 00080975) and operational approval from the regional health authority (AHS # 43638). The results will be disseminated at several levels, including patients, practitioners, academics/researchers, and healthcare organizations.

The investigators will plan an organizational engagement strategy to advance discussions about feasibility and effectiveness prior to the conclusion of the trial. This will help ensure the findings are a relevant part of decision-making processes in a way that is aligned with study findings as they emerge. This may facilitate planning of a larger study that is endorsed at both leadership and operational levels, so that the potential benefits of the interventions can reach patients in a more timely fashion.

DISCUSSION: The results of the study will provide important information about the effectiveness of group CBT and/or group exercise in treatment of MDD. This will augment the literature in this area, and also provide practical benefits in examining if benefit can be derived from group treatment modalities. Currently, patients with MDD referred to AMH Clinics in Edmonton Zone may wait for weeks before receiving care from a health care professional in a one-to-one setting. Long wait may negatively impact patients' well-being, personal and occupational function as well as their satisfaction with care, and a group-based treatment may serve as an alternative for patients with MDD that can be more expediently accessed.

The results of the pilot trial may inform the implementation of a multi-center clinical trial and provide useful information for administrators and clinicians who are interested in incorporating these interventions into existing care. The investigators expect that the pilot findings will inform and support administrative decision-making with respect to further scaling and studying the intervention within the province of Alberta and beyond.

AUTHORS' CONTRIBUTIONS: The study was conceived and designed by VIOA who also contributed to drafting of the initial and final drafts of the manuscript. MH, MYS and GG contributed to the study design and drafting of the initial and final drafts of the manuscript. PC, MS, JM, KD, LL, DT, JK, PC, DS, JC, JB, KH, DL, LF, AD, SD SS and AAA contributed to the study design and revising the initial draft of the of the manuscript. All authors approved of the final draft of the manuscript prior to submission.

FUNDING STATEMENT: This work was supported by a Pfizer Depression grant (via Department of Psychiatry, University of Alberta) and support was received from Alberta Health Services.

COMPETING INTERESTS STATEMENT: All authors have nothing to disclose.

ELIGIBILITY:
Inclusion Criteria:

* Have been referred by a primary care provider or self-referred to the Addiction and Mental Health intake service in Edmonton
* Have received a diagnosis of Major Depressive Disorder from a consultant psychiatrist based on DSM 5 criteria
* Have provided written informed consent

Exclusion Criteria:

* Not meeting the above Inclusion Criteria
* Have not provided informed consent
* Have a diagnosis of Bipolar Disorder, Schizophrenia or Schizoaffective Disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Measuring changes in depressive symptoms scores using Beck Depression Inventory [Symptom Variable - Severity of Depression] | At the enrollment, at the weeks 12 and 24 post enrollment, at the 1st, 7th and 14th week of the 14-week intervention delivery period
  The Beck Depression Inventory (BDI) is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. It contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used are as follows: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
Evaluating change in symptoms using CORE 34 OM [Symptom variable - Symptoms Sub-scale - Psychological Health ] | At the enrollment, at the weeks 12 and 24 post enrollment, at the 1st, 7th and 14th week of the 14-week intervention delivery period
  This is a client self-report questionnaire designed to be administered before and after therapy. The client is asked to respond to 34 questions about how they have been feeling over the last week, using a 5-point scale ranging from 'not at all' to 'most or all of the time'. The questionnaire covers four dimensions: subjective well-being, problems/symptoms, life functioning and risk/harm. Key points in the scoring are as follows: each item within the CORE Outcome Measure is scored on a 5-point scale ranging from 0 (not at all) to 4 (most or all the time). The total score is calculated by adding the response values of all 34 items. The minimum score that can be achieved is 0 and the maximum 136. The total mean score is calculated by dividing the total score by the number of completed item responses. Symptoms sub-scale includes 12 items with a total score range of 0 to 48 and mean score range of 0 to 4 with a cut-off point of 1.44 for males and 1.62 for females.
Evaluating change in risk level using CORE 34 OM [Symptom variable - Risk Sub-scale - Psychological Health ] | At the enrollment, at the weeks 12 and 24 post enrollment, at the 1st, 7th and 14th week of the 14-week intervention delivery period
  This is a client self-report questionnaire designed to be administered before and after therapy. The client is asked to respond to 34 questions about how they have been feeling over the last week, using a 5-point scale ranging from 'not at all' to 'most or all of the time'. The questionnaire covers four dimensions: subjective well-being, problems/symptoms, life functioning and risk/harm. Key points in the scoring are as follows: each item within the CORE Outcome Measure is scored on a 5-point scale ranging from 0 (not at all) to 4 (most or all the time). The total score is calculated by adding the response values of all 34 items. The minimum score that can be achieved is 0 and the maximum 136. The total mean score is calculated by dividing the total score by the number of completed item responses. Risk sub-scale includes 6 items with a total score range of 0 to 24 and mean score range of 0 to 4 with a cut-off point of 0.43 for males and 0.31 for females.
Evaluating change in interpersonal functioning using CORE 34 OM [Functional variable - Functioning Sub-scale - Social Relationship ] | At the enrollment, at the weeks 12 and 24 post enrollment, at the 1st, 7th and 14th week of the 14-week intervention delivery period
  This is a client self-report questionnaire designed to be administered before and after therapy. The client is asked to respond to 34 questions about how they have been feeling over the last week, using a 5-point scale ranging from 'not at all' to 'most or all of the time'. The questionnaire covers four dimensions: subjective well-being, problems/symptoms, life functioning and risk/harm. Key points in the scoring are as follows: each item within the CORE Outcome Measure is scored on a 5-point scale ranging from 0 (not at all) to 4 (most or all the time). The total score is calculated by adding the response values of all 34 items. The minimum score that can be achieved is 0 and the maximum 136. The total mean score is calculated by dividing the total score by the number of completed item responses. Life/ interpersonal functioning sub-scale includes 12 items with a total score range of 0 to 48 and mean score range of 0 to 4 with a cut-off point of 1.29 for males and 1.30 for females.
Evaluating change in well-being using CORE 34 OM [Functional variable - Well-being sub-scale - Psychological Health ] | At the enrollment, at the weeks 12 and 24 post enrollment, at the 1st, 7th and 14th week of the 14-week intervention delivery period
  This is a client self-report questionnaire designed to be administered before and after therapy. The client is asked to respond to 34 questions about how they have been feeling over the last week, using a 5-point scale ranging from 'not at all' to 'most or all of the time'. The questionnaire covers four dimensions: subjective well-being, problems/symptoms, life functioning and risk/harm. Key points in the scoring are as follows: each item within the CORE Outcome Measure is scored on a 5-point scale ranging from 0 (not at all) to 4 (most or all the time). The total score is calculated by adding the response values of all 34 items. The minimum score that can be achieved is 0 and the maximum 136. The total mean score is calculated by dividing the total score by the number of completed item responses. Well-being sub-scale includes 12 items with a total score range of 0 to 48 and mean score range of 0 to 4 with a cut-off point of 1.37 for males and 1.77 for females.
Evaluating change in symptoms, risk level, interpersonal functioning, and well-being using CORE 10 OM [Symptom and Functional Variable - Psychological Health] | At the 1st to 13th week of the 14-week intervention delivery period except week 7 when CORE 34 OM will be administered
  This is a client self-report questionnaire designed to be administered before and after therapy. The client is asked to respond to 10 questions about how they have been feeling over the last week. The questionnaire covers four dimensions: subjective well-being, problems/symptoms, life functioning and risk/harm. Key points in the scoring of the CORE-10 are as follows: Each item is scored on a 5-point scale ranging from 0 ('not at all') to 4 ('most or all the time'). The clinical score is calculated by adding the response values of all 10 items and ranges from 0 to 40. The higher the score the more problems the individual is reporting and/or the more distressed they are. A score of 10 or below denotes a score within the non-clinical range and of 11 or above within the clinical range. Within the clinical range the score of 11 is the lower boundary of the 'mild' level, 15 for the 'moderate' level, and 20 for the 'moderate-to-severe' level. A score of 25 or over marks the 'severe' level.
Change in the level of physical activity using the International Physical Activity Questionnaire [Functional Variable - Physical Activity] | At the enrollment, at the 1st, 7th, and 14th week of the 14-week intervention delivery period
  IPAQ is a self-administered instrument designed for surveillance of physical activity in 15-69 years old adults. It consists of 6 questions and assesses physical activity undertaken across a comprehensive set of domains including walking, moderate-intensity activities and vigorous-intensity activities. Computation of the total score requires summation of the duration (in minutes) and frequency (days) of physical activity. Volume of activity can be computed by weighting each type of activity by its energy requirements defined in METs to yield a score in MET-minutes. METs are multiples of the resting metabolic rate and a MET-minute is computed by multiplying the MET score of an activity by the minutes performed. MET-minute scores are equivalent to kilocalories for a 60 kilogram person. Kilocalories may be computed from MET-minutes using the following equation: MET-min x (weight in kilograms/60 kilograms). MET-minutes/week will be reported.

SECONDARY OUTCOMES:
Evaluating patients satisfaction with the service using Addiction and Mental Health Client Experience Survey [Service variables - Satisfaction with service] | 7 and 14 weeks after commencing the intervention
  The "Addiction and Mental Health Client Experience Survey" is a 25-item self-administered tool gathering client's feedback on their experience with the following domains: 1) intake services, 2) information, communication and education, 3) respecting values, needs and preferences, 4) care plan, 5) coordinating and integrating services, 6) treatment effectiveness, asking them to rate their overall satisfaction with the service (item 22) on a scale of 0 to 10 where 0 stands for "not at all satisfied" and 10 stands for "very satisfied".
Evaluating patients satisfaction with the care and treatment they received using Addiction and Mental Health Client Experience Survey [Service variables - Satisfaction with care and treatment] | 7 and 14 weeks after commencing the intervention
  The "Addiction and Mental Health Client Experience Survey" is a 25-item self-administered tool gathering client's feedback on their experience with the following domains: 1) intake services, 2) information, communication and education, 3) respecting values, needs and preferences, 4) care plan, 5) coordinating and integrating services, 6) treatment effectiveness, asking them to rate the care and treatment they received (item 23) in a scale of 0 to 10 where 0 stands for "worst possible care" and 10 stands for "best possible care".
Number of emergency department presentations in the past 6 months - [Service Variable - Service Utilization] | At the time of enrollment in the study and 6 months after enrollment
  Participant's medical record will be reviewed at two points, at the time of enrollment in the study and 6 months after enrollment, to gather information about their use of health services in the past 6 months. The following data will be extracted: number of emergency department presentations, number of EMS use, number of community Addiction and Mental Health services appointments completed, number of days stayed in inpatient services, number of calls to Crisis and urgent services.
  The aim is to compare pre-post rates within each study arm cohort. Each variable would be analyzed separately to determine differences from pre-study to post-study within each cohort. These data will also be used to determine the probable Social Return on Investment (SROI) of the initiative to the system by showing cost-savings through a decrease/avoidance of service utilization. It will be done by assigning a monetary value to each variable. These values are already endorsed and available.
Number of EMS use in the past 6 months - [Service Variable - Service Utilization] | At the time of enrollment in the study and 6 months after enrollment
  Participant's medical record will be reviewed at two points, at the time of enrollment in the study and 6 months after enrollment, to gather information about their use of health services in the past 6 months. The following data will be extracted: number of emergency department presentations, number of EMS use, number of community Addiction and Mental Health services appointments completed, number of days stayed in inpatient services, number of calls to Crisis and urgent services.
  The aim is to compare pre-post rates within each study arm cohort. Each variable would be analyzed separately to determine differences from pre-study to post-study within each cohort. These data will also be used to determine the probable Social Return on Investment (SROI) of the initiative to the system by showing cost-savings through a decrease/avoidance of service utilization. It will be done by assigning a monetary value to each variable. These values are already endorsed and available.
Number of community Addiction and Mental Health services appointments completed in the past 6 months - [Service Variable - Service Utilization] | At the time of enrollment in the study and 6 months after enrollment
  Participant's medical record will be reviewed at two points, at the time of enrollment in the study and 6 months after enrollment, to gather information about their use of health services in the past 6 months. The following data will be extracted: number of emergency department presentations, number of EMS use, number of community Addiction and Mental Health services appointments completed, number of days stayed in inpatient services, number of calls to Crisis and urgent services.
  The aim is to compare pre-post rates within each study arm cohort. Each variable would be analyzed separately to determine differences from pre-study to post-study within each cohort. These data will also be used to determine the probable Social Return on Investment (SROI) of the initiative to the system by showing cost-savings through a decrease/avoidance of service utilization. It will be done by assigning a monetary value to each variable. These values are already endorsed and available.
Number of days stayed in inpatient services in the past 6 months - [Service Variable - Service Utilization] | At the time of enrollment in the study and 6 months after enrollment
  Participant's medical record will be reviewed at two points, at the time of enrollment in the study and 6 months after enrollment, to gather information about their use of health services in the past 6 months. The following data will be extracted: number of emergency department presentations, number of EMS use, number of community Addiction and Mental Health services appointments completed, number of days stayed in inpatient services, number of calls to Crisis and urgent services.
  The aim is to compare pre-post rates within each study arm cohort. Each variable would be analyzed separately to determine differences from pre-study to post-study within each cohort. These data will also be used to determine the probable Social Return on Investment (SROI) of the initiative to the system by showing cost-savings through a decrease/avoidance of service utilization. It will be done by assigning a monetary value to each variable. These values are already endorsed and available.
Number of calls to Crisis and urgent services in the past 6 months - [Service Variable - Service Utilization] | At the time of enrollment in the study and 6 months after enrollment
  Participant's medical record will be reviewed at two points, at the time of enrollment in the study and 6 months after enrollment, to gather information about their use of health services in the past 6 months. The following data will be extracted: number of emergency department presentations, number of EMS use, number of community Addiction and Mental Health services appointments completed, number of days stayed in inpatient services, number of calls to Crisis and urgent services.
  The aim is to compare pre-post rates within each study arm cohort. Each variable would be analyzed separately to determine differences from pre-study to post-study within each cohort. These data will also be used to determine the probable Social Return on Investment (SROI) of the initiative to the system by showing cost-savings through a decrease/avoidance of service utilization. It will be done by assigning a monetary value to each variable. These values are already endorsed and available.
Social Return on Investment (SROI) of the initiative to the system in the past 6 months - [Service Variable - Service Utilization] | At the time of enrollment in the study and 6 months after enrollment
  Participant's medical record will be reviewed at two points, at the time of enrollment in the study and 6 months after enrollment, to gather information about their use of health services in the past 6 months. The following data will be extracted: number of emergency department presentations, number of EMS use, number of community Addiction and Mental Health services appointments completed, number of days stayed in inpatient services, number of calls to Crisis and urgent services.
  The aim is to compare pre-post rates within each study arm cohort. Each variable would be analyzed separately to determine differences from pre-study to post-study within each cohort. These data will also be used to determine the probable Social Return on Investment (SROI) of the initiative to the system by showing cost-savings through a decrease/avoidance of service utilization. It will be done by assigning a monetary value to each variable. These values are already endorsed and available.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Alexander Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdollahi A, LeBouthillier DM, Najafi M, Asmundson GJG, Hosseinian S, Shahidi S, Carlbring P, Kalhori A, Sadeghi H, Jalili M. Effect of exercise augmentation of cognitive behavioural therapy for the treatment of suicidal ideation and depression. J Affect Disord. 2017 Sep;219:58-63. doi: 10.1016/j.jad.2017.05.012. Epub 2017 May 8. PMID 28525821
- [Background] Bridle C, Spanjers K, Patel S, Atherton NM, Lamb SE. Effect of exercise on depression severity in older people: systematic review and meta-analysis of randomised controlled trials. Br J Psychiatry. 2012 Sep;201(3):180-5. doi: 10.1192/bjp.bp.111.095174. PMID 22945926
- [Background] Catalan-Matamoros D, Gomez-Conesa A, Stubbs B, Vancampfort D. Exercise improves depressive symptoms in older adults: An umbrella review of systematic reviews and meta-analyses. Psychiatry Res. 2016 Oct 30;244:202-9. doi: 10.1016/j.psychres.2016.07.028. Epub 2016 Jul 22. PMID 27494042
- [Background] Cooney G, Dwan K, Mead G. Exercise for depression. JAMA. 2014 Jun 18;311(23):2432-3. doi: 10.1001/jama.2014.4930. PMID 24938566
- [Background] Craft LL, Perna FM. The Benefits of Exercise for the Clinically Depressed. Prim Care Companion J Clin Psychiatry. 2004;6(3):104-111. doi: 10.4088/pcc.v06n0301. PMID 15361924
- [Background] Euteneuer F, Dannehl K, Del Rey A, Engler H, Schedlowski M, Rief W. Immunological effects of behavioral activation with exercise in major depression: an exploratory randomized controlled trial. Transl Psychiatry. 2017 May 16;7(5):e1132. doi: 10.1038/tp.2017.76. PMID 28509904
- [Background] Gill A, Womack R, Safranek S. Clinical Inquiries: Does exercise alleviate symptoms of depression? J Fam Pract. 2010 Sep;59(9):530-1. PMID 20824231
- [Background] Huang TT, Liu CB, Tsai YH, Chin YF, Wong CH. Physical fitness exercise versus cognitive behavior therapy on reducing the depressive symptoms among community-dwelling elderly adults: A randomized controlled trial. Int J Nurs Stud. 2015 Oct;52(10):1542-52. doi: 10.1016/j.ijnurstu.2015.05.013. Epub 2015 Jun 10. PMID 26105535
- [Background] Josefsson T, Lindwall M, Archer T. Physical exercise intervention in depressive disorders: meta-analysis and systematic review. Scand J Med Sci Sports. 2014 Apr;24(2):259-72. doi: 10.1111/sms.12050. Epub 2013 Jan 30. PMID 23362828
- [Background] Mead GE, Morley W, Campbell P, Greig CA, McMurdo M, Lawlor DA. Exercise for depression. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD004366. doi: 10.1002/14651858.CD004366.pub4. PMID 19588354
- [Background] Schuch FB, Vancampfort D, Richards J, Rosenbaum S, Ward PB, Stubbs B. Exercise as a treatment for depression: A meta-analysis adjusting for publication bias. J Psychiatr Res. 2016 Jun;77:42-51. doi: 10.1016/j.jpsychires.2016.02.023. Epub 2016 Mar 4. PMID 26978184
- [Derived] Yekrang Safakar M, Hrabok M, Urichuk L, Juhas M, Shalaby R, Parmar D, Chue P, Snaterse M, Mason J, Tchida D, Kelland J, Coulson P, Sosdjan D, Brown J, Hay K, Lesage D, Paulsen L, Delday A, Duiker S, Surood S, Abba-Aji A, Agyapong VIO. Effectiveness of Group Cognitive Behavioral Therapy and Exercise in the Management of Major Depressive Disorder: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2020 May 25;9(5):e14309. doi: 10.2196/14309. PMID 32449684
- See also: Depression and other common mental disorders: global health estimates. — http://apps.who.int/iris/bitstream/handle/10665/254610/WHO-MSD-MER-2017.2-eng.pdf
- See also: Depression in adults: recognition and management | Guidance and guidelines | NICE — https://www.nice.org.uk/guidance/cg90
- See also: Edmonton, C. of. (2017, September 14). 2016 Municipal Census Results. — https://www.edmonton.ca/city_government/facts_figures/municipal-census-results.aspx

DOCUMENTS (2):
  • Study Protocol (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03731728/Prot_002.pdf
  • Informed Consent Form (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03731728/ICF_003.pdf